CLINICAL TRIAL: NCT03330431
Title: Effects of Videos Aiming to Optimize Expectations on Effectiveness of Progressive Muscle Relaxation (PMR)
Brief Title: Do Videos That Aim to Optimize Expectations Alter the Effectivess of PMR?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Winfried Rief, Prof. Dr., Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017_EXPECT_v1
Record Dates: First submitted 2017-09-27; First posted 2017-11-06 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: Experimental Group 1 (Video Personal Expert); Experimental Group 2 (Video Factual Expert); Control Group
MeSH Terms: interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 1 (personal expert) (Experimental): Participants watch a video of an expert describing the positive effects of Progressive Muscle Relaxation (PMR) with personalized examples and stories before undergoing a PMR session.
  Interventions: Behavioral: Progressive Muscle Relaxation (PMR)
- Experimental group 2 (factual expert) (Experimental): Participants watch a video of an expert describing the positive effects of Progressive Muscle Relaxation (PMR) with factual information (not personal) before undergoing a PMR session.
  Interventions: Behavioral: Progressive Muscle Relaxation (PMR)
- Control group (Active Comparator): Participants read a neutral text before undergoing a Progressive Muscle Relaxation (PMR) session.
  Interventions: Behavioral: Progressive Muscle Relaxation (PMR)

INTERVENTIONS:
Behavioral: Progressive Muscle Relaxation (PMR) — All groups undergo a PMR session, but they differ regarding the treatment before the PMR session. Two groups watch a video before undergoing PMR, the control group reads a text before undergoing PMR.
  Progressive muscle relaxation (PMR) is a technique for learning to monitor and control the state of muscular tension. It was developed by American physician Edmund Jacobson in the early 1920s.
  The technique involves learning to monitor tension in each specific muscle group in the body by deliberately inducing tension in each group. This tension is then released, with attention paid to the contrast between tension and relaxation.

SUMMARY:
The study's aim is to determine whether a short video aiming to optimize expectations regarding the effectiveness of progressive muscle relaxation (PMR) ist able to improve the actual effectiveness of PMR in comparison with a neutral (no video) control group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants
* fluency in the German language to provide informed consent

Exclusion Criteria:

* Chronic illness
* Mental disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Change in perceived/subjective relaxation | Change from pre (baseline) to post scores (30 minutes later)
  Participants are asked to rate how relaxed they feel at the moment at two time points (baseline and after the PMR intervention) on a questionnaire (VAS: item ranges from 0 (not relaxed at all) - 100 (very relaxed). Change scores are calculated (post- minus pre-scores).

SECONDARY OUTCOMES:
Change in perceived stress | Change from pre (baseline) to post scores (30 minutes later)
  Participants are asked to rate how stressed they feel at the moment at two time points (baseline and after the PMR intervention) on a questionnaire (VAS: item ranges from 0 (not stressed at all) - 100 (very stressed). Change scores are calculated (post- minus pre-scores).
Change in physiological relaxation | Change from pre (baseline) to post scores (30 minutes later)
  Electromyography is used to assess participants' physiological relaxation status at baseline and after the PMR intervention. Change scores are calculated (post- minus pre-scores).

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Professor, Principal Investigator — Philipps Universität Marburg
Locations (1):
- Department of Psychology, Philipps University Marburg, Marburg, Hesse, Germany

REFERENCES:
- [Derived] Salzmann S, Wilhelm M, Schindler S, Rief W, Euteneuer F. Optimising the efficacy of a stress-reducing psychological intervention using placebo mechanisms: A randomized controlled trial. Stress Health. 2022 Oct;38(4):722-735. doi: 10.1002/smi.3128. Epub 2022 Jan 24. PMID 35043534